CLINICAL TRIAL: NCT06463665
Title: A Randomized Phase 2 Study Assessing the Efficacy and Safety of Olvimulogene Nanivacirepvec Followed by Platinum-doublet Chemotherapy + Physician's Choice of Immune Checkpoint Inhibitor Compared With Docetaxel in Patients With NSCL Cancer After First Progression While on Front-line Immune Checkpoint Inhibitor-based Maintenance
Brief Title: Efficacy & Safety of Olvimulogene Nanivacirepvec & Platinum-doublet + Physician's Choice of Immune Checkpoint Inhibitor Compared to Docetaxel in NSCL Cancer
Acronym: VIRO-25
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genelux Corporation (Industry)
Collaborators: Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Olvi-Vec-NSCLC-025
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Advanced Non-squamous Non-small-cell Lung Cancer; Advanced Squamous Non-Small Cell Lung Carcinoma; Metastatic Non-squamous Non Small Cell Lung Cancer; Metastatic Squamous Non-Small Cell Lung Carcinoma; Non-small Cell Lung Cancer; Non-small Cell Lung Cancer Stage III; Non-small Cell Lung Cancer Stage IV; Non-small Cell Lung Cancer Recurrent
Keywords: Olvi-Vec; virotherapy; viral therapy; immunotherapy; immunochemotherapy; combination therapy; vaccinia virus; platinum-doublet chemotherapy; pembrolizumab; nivolumab; cemiplimab; atezolizumab; durvalumab; anti-PD-1; anti-PD-L1; carboplatin; cisplatin; docetaxel; neoplasms by site; neoplasms; carcinoma; Neoplasms by Histologic type; Antineoplastic Agents, Phytogenic; Antineoplastic Agents; Antimitotic Agents; Molecular Mechanisms of Pharmacological Action; Immune Checkpoint Inhibitors; NSCLC; NSCL cancer; chemoimmunotherapy; ICI; platinum resensitization; platinum resistant; chemoresistance; resensitize; olvimulogene nanivacirepvec
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Vaccinia; Neoplasms by Site; Neoplasms; Carcinoma; Neoplasms by Histologic Type | interventions — Cisplatin; 130-nm albumin-bound paclitaxel; Pemetrexed; Nivolumab; cemiplimab; atezolizumab; durvalumab; Docetaxel

STUDY DESIGN:
Intervention Model Description: Following selection of the dose and schedule from the three safety run-in cohorts, randomization is (1:1) either into the Experimental Arm (EA) which is Olvi-Vec with platinum-doublet + Physician's Choice of ICI and then ICI-based maintenance or in the Active Comparator Arm (ACA) which includes treatment with docetaxel. ACA patients with documented disease progression [i.e., assessed by Blinded Independent Central Review (BICR)] who are eligible may crossover to receive the same treatment as per the Experimental Arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single-arm run-in Olvi-Vec dose escalation Cohorts (Experimental): Cohort 1: Olvi-Vec administered over 3 consecutive days at 0.5,0.5,0.5 x 10e9 pfu followed 2 to 3 weeks later with platinum-doublet chemotherapy + Physician's Choice of ICI.
  Cohort 2: Olvi-Vec administered over 3 consecutive days at 1,1,1 x 10e9 pfu followed 2 to 3 weeks later with platinum-doublet chemotherapy + Physician's Choice of ICI.
  Cohort 3: Olvi-Vec administered over 4 consecutive days at 1,2,3 x 10e9 pfu followed 2 to 3 weeks later with platinum-doublet chemotherapy + Physician's Choice of ICI.
  Interventions: Biological: Olvimulogene nanivacirepvec; Drug: Platinum chemotherapy: carboplatin or cisplatin; Drug: Non-platinum chemotherapy: paclitaxel or nab-paclitaxel for squamous cell NSCLC or pemetrexed for nonsquamous cell NSCLC; Drug: Physician's Choice of Immune Checkpoint Inhibitor: pembrolizumab, nivolumab, cemiplimab, atezolizumab, durvalumab
- Experimental Arm (Experimental): Olvi-Vec will be administered at the dose and schedule selected from the single-arm run-in Olvi-Vec dose escalation cohorts followed 2 to 3 weeks later with platinum-doublet chemotherapy + Physician's Choice of ICI.
  Interventions: Biological: Olvimulogene nanivacirepvec; Drug: Platinum chemotherapy: carboplatin or cisplatin; Drug: Non-platinum chemotherapy: paclitaxel or nab-paclitaxel for squamous cell NSCLC or pemetrexed for nonsquamous cell NSCLC; Drug: Physician's Choice of Immune Checkpoint Inhibitor: pembrolizumab, nivolumab, cemiplimab, atezolizumab, durvalumab
- Active Comparator Arm (Active Comparator): Docetaxel starts in Week 0 and continues until disease progression is assessed by the BICR.
  Interventions: Drug: Docetaxel
- Active Comparator Arm Cross-over (Other): Patients randomized into the Active Comparator can cross-over to receive the same treatment as given in the Experimental Arm following determination of (1) disease progression by BICR after receiving docetaxel treatment and (2) confirming eligibility.
  Interventions: Biological: Olvimulogene nanivacirepvec; Drug: Platinum chemotherapy: carboplatin or cisplatin; Drug: Non-platinum chemotherapy: paclitaxel or nab-paclitaxel for squamous cell NSCLC or pemetrexed for nonsquamous cell NSCLC; Drug: Physician's Choice of Immune Checkpoint Inhibitor: pembrolizumab, nivolumab, cemiplimab, atezolizumab, durvalumab; Drug: Docetaxel

INTERVENTIONS:
Biological: Olvimulogene nanivacirepvec — Olvi-Vec is an engineered oncolytic vaccinia virus
  Other Names: Olvi-Vec; GL-ONC; GLV-1h68
  Arms: Active Comparator Arm Cross-over; Experimental Arm; Single-arm run-in Olvi-Vec dose escalation Cohorts
Drug: Platinum chemotherapy: carboplatin or cisplatin — Administered according to local practice.
  Other Names: Brand of drug is based on institutional procurement
  Arms: Active Comparator Arm Cross-over; Experimental Arm; Single-arm run-in Olvi-Vec dose escalation Cohorts
Drug: Non-platinum chemotherapy: paclitaxel or nab-paclitaxel for squamous cell NSCLC or pemetrexed for nonsquamous cell NSCLC — Administered according to local practice.
  Other Names: Brand of drug is based on institutional procurement
  Arms: Active Comparator Arm Cross-over; Experimental Arm; Single-arm run-in Olvi-Vec dose escalation Cohorts
Drug: Physician's Choice of Immune Checkpoint Inhibitor: pembrolizumab, nivolumab, cemiplimab, atezolizumab, durvalumab — Administered according to local practice.
  Other Names: Brand of drug is based on institutional procurement
  Arms: Active Comparator Arm Cross-over; Experimental Arm; Single-arm run-in Olvi-Vec dose escalation Cohorts
Drug: Docetaxel — Administered according to local practice.
  Other Names: Brand of drug is based on institutional procurement
  Arms: Active Comparator Arm; Active Comparator Arm Cross-over

SUMMARY:
This Phase 2, open-label, randomized study in non-small-cell lung cancer (NSCLC) is designed to evaluate the efficacy and safety of an intravenously delivered oncolytic vaccinia virus, Olvi-Vec, followed by platinum-doublet chemotherapy + Physician's Choice of Immune Checkpoint Inhibitor (ICI) vs. docetaxel for patients with advanced or metastatic NSCLC who have shown first disease progression (i.e., progressive disease not yet confirmed by further scan after initial scan showing progression) while on front-line treatment or maintenance ICI therapy after front-line treatment with platinum-doublet chemotherapy + ICI as standard of care.

DETAILED DESCRIPTION:
Olvi-Vec (olvimulogene nanivacirepvec, aka GL-ONC1; laboratory name: GLV-1h68) is an oncolytic vaccinia virus-based immunotherapy that has been shown to have broad infectivity in a wide range of tumor types including non-small-cell lung cancer (NSCLC). In preclinical studies, Olvi-Vec was shown to infect and kill NSCLC cells and tumors in vitro and in vivo, respectively, and resolved and prevented formation of malignant effusion. This study is to test the hypothesis that the combination of Olvi-Vec followed by further platinum-based chemotherapy plus an ICI is particularly effective against established tumors by virus-mediated immune activation and re-sensitization of tumor cells to chemotherapy. Participants will have advanced or metastatic NSCLC (Stage III or Stage IV) squamous or nonsquamous disease without known targetable alterations in Epidermal Growth Factor Receptor (EGFR), Anaplastic Lymphoma Kinase (ALK) or Repressor of Silencing 1 (ROS1). Eligible patients will have first disease progression by radiological assessment (i) while on front-line platinum-doublet chemotherapy and ICI, or (ii) while receiving front-line maintenance ICI-based therapy after completion of front-line therapy, with at least 2 cycles and maximum of 6 cycles of platinum-doublet chemotherapy and ICI, regardless of Programmed death-ligand 1 (PD-L1) expression as the first treatment after being diagnosed. ICI includes anti-programmed death-1 (anti-PD-1) or anti-PD-L1 agents. Other classes of ICI [e.g., anti-cytotoxic T-lymphocyte antigen 4 (anti-CTLA-4), etc.] are excluded. Patients will be stratified based on length of time on ICI-based therapy from start date of the first dose, if ICI during front-line therapy, until date of first progression by radiological assessment is either less than or equal to 4 months or greater than 4 months. Patients enrolled in one of the initial 3 cohorts will receive either 3 or 4 days of Olvi-Vec followed by platinum-doublet chemotherapy + Physician's Choice of ICI. The randomization part of the study will start afterwards with the Olvi-Vec dose and schedule selected from one of the 3 cohorts for the Experimental Arm. The Active Comparator Arm (ACA) treatment includes docetaxel. Participants treated in the ACA who subsequently have documented disease progression may cross-over for treatment as per the Experimental Arm following determination of eligibility.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.
* Have histologically or cytologically confirmed advanced or metastatic NSCLC.
* Histologically confirmed Stage III or IV squamous or nonsquamous [American Joint Committee on Cancer (AJCC) 8th edition].
* Received at least 2 cycles and maximum of 6 cycles of front-line platinum-based chemotherapy with ICI-based therapy, regardless of PD-L1 expression.
* Reached first disease progression by radiological assessment while receiving front-line or maintenance ICI.
* At least one measurable target tumor lesion anywhere except the brain per RECIST 1.1 by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scan.
* Have adequate renal, hepatic, bone marrow function as well as adequate coagulation tests [International Normalized Ratio (INR)] and adequate immune function by lymphocyte count.
* Women of child-bearing potential must have a negative serum pregnancy test prior to initiating study dosing.
* Be willing and able to comply with scheduled visits, the treatment plan, imaging and laboratory tests.

Exclusion Criteria:

* Active and untreated urinary tract infection, pneumonia, or other systemic infections.
* Current symptomatic central nervous system (CNS) metastasis.
* Any uncontrolled systemic disease, condition or comorbidity that, in the opinion of the Investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Persistent toxicities [Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 3] caused by previous anticancer therapy; alopecia and vitiligo are excluded toxicities.
* Required the use of additional immunosuppression other than corticosteroids for the management of an adverse event or have experienced recurrence of an adverse event if re-challenged, or currently require maintenance doses of >10 mg prednisone or equivalent per day.
* Receiving concurrent antiviral agent active against vaccinia virus (e.g., cidofovir, vaccinia immunoglobulin, imatinib, tecovirimat, or other agents with known anti-vaccinia activities).
* Underwent major surgery within 4 weeks, or have insufficient recovery from surgical-related trauma or wound healing, prior to the planned first dose of treatment in either Arm.
* Have received prior virus-based gene therapy or therapy with cytolytic virus of any type.
* Vaccination against smallpox or monkeypox within 1 year of study therapy.
* Any non-oncology vaccine therapy used for prevention of infectious diseases, such as seasonal (influenza) vaccinations, corona virus disease (COVID) vaccination or other vaccines, within 2 weeks of the planned first dose of study drug.
* Clinically significant skin disease as assessed by the Investigator (e.g., severe eczema, psoriasis, or any unresolved skin injury or ulcer).
* Known hypersensitivity to carboplatin, cisplatin, paclitaxel or nab-paclitaxel, docetaxel, or any of the constituents of Olvi-Vec (i.e., gentamicin).
* Had severe hypersensitivity (CTCAE Grade ≥ 3) to ICI and/or any of its excipients previously.
* Dementia or altered mental status that would prohibit informed consent, and/or psychiatric illness/social situations that might interfere or limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Blinded Independent Central Review (BICR) | From date of randomization up to 12 months.
  To assess progression-free survival from time of randomization until first documented disease progression based on radiological assessment or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by RECIST 1.1 | From date of randomization up to 12 months.
  Ratio of the sum of complete responses (CR) & partial responses (PR) divided by the number of participants from start of treatment to confirmation of response.
Median Overall Survival | From date of randomization up to 36 months.
  Time from randomization until death or study completion; assessed up to 36 months.
Six-month Progression-free Survival Rate | From date of randomization up to 6 months.
  Proportion of patients who remained alive and progression-free at 6 months.
Incidence of Treatment-emergent Adverse Events | Assessed up to 36 months.
  From date of first study treatment until death or study completion.
Duration of Response by RECIST 1.1 | From date of randomization up to 12 months.
  Time from date of first response until the first date of progressive disease based on radiological assessment.
Disease Control Rate (DCR) | From date of randomization up to 12 months.
  Percentage of patients who have achieved complete response, partial response or stable disease out of the total number of patients evaluated in a therapeutic intervention in clinical trials: DCR = [CR + PR + SD (stable disease)]/total # of patients evaluated by RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Pioneer Research Center, LLC, Bullhead City, Arizona
  - Clermont Oncology Center, Clermont, Florida
  - Oncology & Hematology Associates of West Broward, Coral Springs, Florida
  - Helios Clinical Research, Fort Lauderdale, Florida
  - Bioresearch Partner, Hialeah, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Bioresearch Partner, Miami, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - BRCR Medical Center, Inc., Plantation, Florida
  - University of Maryland Medical Center Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Michigan Hematology and Oncology Consultants, Dearborn, Michigan
  - Oakland Medical Group, Farmington Hills, Michigan
  - Gabrail Cancer and Research Center, Canton, Ohio
  - Texas Oncology - Austin Central, Austin, Texas
  - World Research Link, Baytown, Texas
  - Sheboygan Cancer & Blood Center, Sheboygan, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's website — http://www.genelux.com